CLINICAL TRIAL: NCT05988099
Title: Comparison of the Effects of Standardized Chokeberry Extracts With Various Formulations on the Levels of Selected Markers Associated With Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 04-AP-MEL
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Hypertension; Hypercholesterolemia
Keywords: Hypertension; Hypercholesterolemia; Aronia extract; Chokeberry extract
MeSH Terms: conditions — Hypertension; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Complex product (chokeberry extract, L-arginine, vitamin E, vitamin A, folic acid, chromium) (Experimental): Single oral dose - 2 capsules
  Interventions: Dietary Supplement: Complex product
- Chokeberry extract in liposomal formulation (Active Comparator): Single oral dose - 2 capsules
  Interventions: Dietary Supplement: Chokeberry extract in liposomal formulation
- Chokeberry extract in traditional formulation (Active Comparator): Single oral dose - 2 capsules
  Interventions: Dietary Supplement: Chokeberry extract in traditional formulation
- Placebo (Placebo Comparator): Single oral dose - 2 capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Complex product — 400 mg of chokeberry extract in liposomal formulation and L-arginine, vitamin E, vitamin A, folic acid, chromium
  Arms: Complex product (chokeberry extract, L-arginine, vitamin E, vitamin A, folic acid, chromium)
Dietary Supplement: Chokeberry extract in liposomal formulation — 400 mg of chokeberry extract in liposomal formulation
  Arms: Chokeberry extract in liposomal formulation
Dietary Supplement: Chokeberry extract in traditional formulation — 400 mg of chokeberry extract in traditional formulation
  Arms: Chokeberry extract in traditional formulation
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to compare in a clinical condition the effect of standardized chokeberry extract in different formulations and a complex preparation containing chokeberry extract and other active ingredients in on the levels of selected markers associated with cardiovascular diseases in people with a predisposition to the development of these diseases.

DETAILED DESCRIPTION:
Randomized, double-blind, parallel study conducted under medical supervision on a group of 40 patients with known hypertension and/or hypercholesterolemia. Patients receive one of the investigational products or placebo for 6 weeks. Before and after the study, the following parameters are analyzed: extended lipid panel (total cholesterol (TC), triglycerides (TG), low-density lipoprotein (LDL), HDL and lipoprotein A, apolipoprotein Apo A1 and Apo B), levels of glucose, insulin, homocysteine, markers of kidney and liver function (alanine aminotransferase (ALT), aspartate aminotransferase (AST), lactate dehydrogenase (LDH), blood urea nitrogen (BUN), uric acid). Effects on blood pressure and anthropometric parameters are also being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18-55 years old
* Patients with known: hypertension or hypercholesterolemia,
* Patients on hypotensive or hypolipemic therapy for at least 6 months prior to study enrollment
* Signed informed consent

Exclusion Criteria:

* Intake of supplements containing plant extracts, polyphenols or anthocyanins,
* Intake of supplements with antioxidant properties,
* Participation in another clinical trial,
* Women who are pregnant, planning to become pregnant during the study, or breastfeeding,
* Oncological disease, autoimmune disease, severe liver dysfunction, tuberculosis, leukemia, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplant,
* Patients receiving glucocorticosteroids, anti-allergic drugs, non-steroidal anti-inflammatory drugs in exacerbations of chronic disease.
* Patients with signs of inflammation such as increased body temperature, redness, swelling, pain.
* Patients who have not given written consent to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Extended lipid panel (total cholesterol (TC), triglycerides (TG), low-density lipoprotein (LDL), HDL and lipoprotein A, apolipoprotein Apo A1 and Apo B) | baseline, 6 weeks
  Comparison of lipid panel markers
Glucose level | baseline, 6 weeks
  Comparison of glucose level
Systolic, diatolic blood pressure | baseline, 6 weeks
  Comparison of blood pressure

SECONDARY OUTCOMES:
Insulin level | baseline, 6 weeks
  Comparison of insulin level
Homocysteine level | baseline, 6 weeks
  Comparison of homocysteine level
Alanine aminotransferase (ALT), aspartate aminotransferase (AST) | baseline, 6 weeks
  Comparison of ALT and AST

CONTACTS AND LOCATIONS:
Locations (1):
- Centum Zdrowia Eter-Med sp. z o.o., Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No